CLINICAL TRIAL: NCT03821090
Title: A Study in Subclinical Atherosclerosis in Patients With Rheumatoid Arthritis
Brief Title: Rheumatoid Arthritis Disease Activity and Sub Clinical Atherosclerosis
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sabrin Refaat Mahmoud, principle investigator, Assiut University
Other Study IDs: cardiac affection in RA
Record Dates: First submitted 2019-01-27; First posted 2019-01-29 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: Eighty rheumatoid arthritis patients fulfilling American College of Rheumatology (ACR) 2010 classification criteria, all of them will be subjected to
  1. History including disease duration , course and associated diseases
  2. Clinical examination with specific joint examination
  3. RA disease activity will be evaluated by a 28- joint DAS (DAS28). 4-12-lead ECG
  5-Echocardiography 6-Carotid intima media thickness using carotid doppler 7-Venous blood will be withdrawn to do the following laboratory tests
  1. Complete Blood Count(CBC)
  2. Erythrocyte Sedimentation Rate (ESR) &C Reactive Protein(CRP)
  3. Rheumatoid Factor (RF)& anti cyclic citrullinated peptide (Anti-CCP)
  4. Urine analysis , Urea and creatinine ,
  5. Uric acid level
  6. Lipogram
  7. HA1C
  8. TNF α
  9. hs-cTnI
- control: Eighty healthy subjects age and sex matched will be included , all of them will be subjected to
  1. History
  2. Clinical examination . 3-12-lead ECG
  4-Echocardiography 5-Carotid intima media thickness using carotid doppler 6-Venous blood will be withdrawn to do the following laboratory tests
  1. Complete Blood Count (CBC)
  2. ESR & CRP
  3. RF& Anti-CCP
  4. Urine analysis , Urea and creatinine
  5. Uric acid level
  6. Lipogram
  7. HA1C
  8. TNF α
  9. hs-cTnI

SUMMARY:
RA is associated with traditional cerebrovascular risk factors as subclinical atherosclerosis.

Chronic inflammation and high disease activity are associated with atherosclerotic burden, higher incidence of cerebrovascular disease ,chronic heart failure , and mortality of patients with RA .

High-sensitivity cardiac troponin I (hs-cTnI) predicted a greater risk coronary heart disease, heart failure hospitalization and overall mortality in the general population .

So the aim of the study is to correlate between high sensitive cardiac troponin I , TNF-α to disease activity and presence of subclinical atherosclerosis in RA patients

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory autoimmune disease characterized by progressive joint destruction, associated with extra-articular manifestations, affecting different internal organs .

Interestingly, these patients show an increased risk of mortality when compared to general population and recent evidence clearly confirmed that this risk is largely due to cerebro-cardiovascular events (CV Es), this may be explained by the greater prevalence, severity, burden and different composition of occult coronary lesions in RA compared with age- and gender-matched controls.

RA is associated with traditional CV risk factors ,subclinical atherosclerosis,arrhythmias , and coronary calcifications .

Increased subclinical atherosclerosis, mainly carotid artery plaques, may be observed in RA patients, the increased carotid intima-media thickness (cIMT) and presence of plaques are accepted as strong predictors of generalized atherosclerosis and major CVEs in both non-RA and RA subjects.

The evidence of traditional CV risk factors and subclinical atherosclerosis does not fully explain the increased incidence of CVEs in these patients; suggesting that the CV risk may be independently associated with RA and in fact, this risk has been shown to be associated with additional features specific of RA, such as the systemic inflammatory process, disease duration and therapeutic strategies .

Chronic inflammation and high disease activity are reportedly associated with atherosclerotic burden, higher incidence of cerebrovascular disease (CVD), chronic heart failure (CHF), and mortality of patients with RA . Residual disease activity may further associate with more advanced, complex and prone-to-rupture coronary plaques .

Pro-inflammatory cytokines such as tumor necrosis factor alpha (TNF-α), reflect clinical activity and structural damage in RA and are elevated in the blood of RA patients compared with controls , the same cytokine have been identified in atherosclerotic plaque and correlated with subclinical atherosclerosis independent of cardiac risk factors coronary plaque complexity , plaque destabilization and CVEs in subjects without autoimmune disease .

Cardiac troponins (cTn) are components of the cardiomyocyte contractile apparatus, and circulating concentrations are elevated in the setting of myocardial injury, such as acute coronary syndromes (ACS) .

High-sensitivity (hs) cTn assays allow measurement of troponin concentrations below conventional levels of detection and have revealed a spectrum of circulating cTn concentrations spanning low and high levels in both healthy subjects and in patients with overt cardiovascular disease

Additionally, both high-sensitivity cardiac troponin T (hs-cTnT) and high-sensitivity cardiac troponin I (hs-cTnI) predicted a greater risk of fatal and non-fatal coronary heart disease, heart failure hospitalization and overall mortality in the general population .

Aim of the study

1. Detection of subclinical atherosclerosis in RA patients by means of carotid Doppler
2. Detection of levels of high sensitive cardiac troponin I and TNF-α in RA patients
3. Correlation between high sensitive cardiac troponin I and TNF- α to disease activity and to the presence of subclinical atherosclerosis in RA patients

ELIGIBILITY:
Inclusion Criteria:

* RA patients fulfilling ACR 2010 classification criteria over the age of 18 who have active RA (either early with symptoms lasting < 6 months or established disease lasting > 6 months) .

Exclusion Criteria:

Patients who have previously experienced cardiovascular illness, e.g., heart failure, acute coronary syndrome, revascularization, transient ischemic attacks, and cerebrovascular stroke. Patients who have concomitant hepatic or renal diseases, active infections, malignancy, smoking, hypertension, dyslipidemia, obesity, diabetes mellitus, and hyperuricemia. Patients who are receiving anti-TNF-α therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eighty rheumatoid arthritis patients fulfilling ACR 2010 classification criteria will be in rolled in the study also eighty healthy subjects age and sex matched will be included .
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
detection of subclinical atherosclerosis in RA patients who have no cardiovascular risk factors | baseline
  Correlation between high sensitive cardiac troponin I and TNF- α to disease activity and presence of subclinical atherosclerosis in RA patients

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambrosino P, Lupoli R, Di Minno A, Tasso M, Peluso R, Di Minno MN. Subclinical atherosclerosis in patients with rheumatoid arthritis. A meta-analysis of literature studies. Thromb Haemost. 2015 May;113(5):916-30. doi: 10.1160/TH14-11-0921. Epub 2015 Feb 26. PMID 25716931
- [Background] Baghdadi LR, Woodman RJ, Shanahan EM, Mangoni AA. The impact of traditional cardiovascular risk factors on cardiovascular outcomes in patients with rheumatoid arthritis: a systematic review and meta-analysis. PLoS One. 2015 Feb 17;10(2):e0117952. doi: 10.1371/journal.pone.0117952. eCollection 2015. PMID 25689371
- [Background] Amar J, Fauvel J, Drouet L, Ruidavets JB, Perret B, Chamontin B, Boccalon H, Ferrieres J. Interleukin 6 is associated with subclinical atherosclerosis: a link with soluble intercellular adhesion molecule 1. J Hypertens. 2006 Jun;24(6):1083-8. doi: 10.1097/01.hjh.0000226198.44181.0c. PMID 16685208
- [Background] Bradham WS, Bian A, Oeser A, Gebretsadik T, Shintani A, Solus J, Estis J, Lu QA, Todd J, Raggi P, Stein CM. High-sensitivity cardiac troponin-I is elevated in patients with rheumatoid arthritis, independent of cardiovascular risk factors and inflammation. PLoS One. 2012;7(6):e38930. doi: 10.1371/journal.pone.0038930. Epub 2012 Jun 28. PMID 22761714
- [Background] deFilippi CR, de Lemos JA, Christenson RH, Gottdiener JS, Kop WJ, Zhan M, Seliger SL. Association of serial measures of cardiac troponin T using a sensitive assay with incident heart failure and cardiovascular mortality in older adults. JAMA. 2010 Dec 8;304(22):2494-502. doi: 10.1001/jama.2010.1708. Epub 2010 Nov 15. PMID 21078811
- [Background] Gupta S, de Lemos JA. Use and misuse of cardiac troponins in clinical practice. Prog Cardiovasc Dis. 2007 Sep-Oct;50(2):151-65. doi: 10.1016/j.pcad.2007.01.002. PMID 17765476
- [Background] Karpouzas GA, Malpeso J, Choi TY, Li D, Munoz S, Budoff MJ. Prevalence, extent and composition of coronary plaque in patients with rheumatoid arthritis without symptoms or prior diagnosis of coronary artery disease. Ann Rheum Dis. 2014 Oct;73(10):1797-804. doi: 10.1136/annrheumdis-2013-203617. Epub 2013 Jul 25. PMID 23887286
- [Background] Lazzerini PE, Capecchi PL, Acampa M, Galeazzi M, Laghi-Pasini F. Arrhythmic risk in rheumatoid arthritis: the driving role of systemic inflammation. Autoimmun Rev. 2014 Sep;13(9):936-44. doi: 10.1016/j.autrev.2014.05.007. Epub 2014 May 27. PMID 24874445
- [Background] Fransen J, Kazemi-Bajestani SM, Bredie SJ, Popa CD. Rheumatoid Arthritis Disadvantages Younger Patients for Cardiovascular Diseases: A Meta-Analysis. PLoS One. 2016 Jun 16;11(6):e0157360. doi: 10.1371/journal.pone.0157360. eCollection 2016. PMID 27310259
- [Background] McInnes IB, Schett G. The pathogenesis of rheumatoid arthritis. N Engl J Med. 2011 Dec 8;365(23):2205-19. doi: 10.1056/NEJMra1004965. No abstract available. PMID 22150039
- [Background] Navarro-Millan I, Yang S, DuVall SL, Chen L, Baddley J, Cannon GW, Delzell ES, Zhang J, Safford MM, Patkar NM, Mikuls TR, Singh JA, Curtis JR. Association of hyperlipidaemia, inflammation and serological status and coronary heart disease among patients with rheumatoid arthritis: data from the National Veterans Health Administration. Ann Rheum Dis. 2016 Feb;75(2):341-7. doi: 10.1136/annrheumdis-2013-204987. Epub 2015 Jan 21. PMID 25609412
- [Background] Niemann-Jonsson A, Dimayuga P, Jovinge S, Calara F, Ares MP, Fredrikson GN, Nilsson J. Accumulation of LDL in rat arteries is associated with activation of tumor necrosis factor-alpha expression. Arterioscler Thromb Vasc Biol. 2000 Oct;20(10):2205-11. doi: 10.1161/01.atv.20.10.2205. PMID 11031205